CLINICAL TRIAL: NCT07015671
Title: Bioavailability and Bioequivalence (BA/BE) Study of Extended Release (ER) Torsemide and Spironolactone Fixed Dose Combination (FDC) Tablet in Healthy Subjects
Brief Title: Bioavailability and Bioequivalence Study of ER Torsemide and Spironolactone FDC Tablet in Healthy Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAR-HS-025-23
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Bioequivalence Study in Healthy Subjects; PK/PD
Keywords: torsemide; Spironolactone; bioequivalence; diuresis; extended release; immediate release; PK/PD
MeSH Terms: interventions — Torsemide; Spironolactone; Tablets

STUDY DESIGN:
Intervention Model Description: Open label, randomized, four period, four sequence, balanced, single dose, crossover BA/BE study of the fixed dose combination (FDC) and its components administered individually or together, under fasting conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): 10 mg Torsemide tablet
  Interventions: Drug: 10 mg Torsemide tablet
- Treatment B (Experimental): 25 mg Aldactone (Spironolactone) tablet
  Interventions: Drug: 25 mg Aldactone (Spironolactone) tablet
- Treatment C (Experimental): FDC (12 mg ER Torsemide + 15 mg Spironolactone) tablet
  Interventions: Drug: FDC (12 mg ER Torsemide + 15mg Spironolactone) tablet
- Treatment D (Experimental): 10 mg Torsemide tablet and 25 mg Aldactone® (Spironolactone) tablet given together
  Interventions: Drug: 10 mg Torsemide tablet; Drug: 25 mg Aldactone (Spironolactone) tablet

INTERVENTIONS:
Drug: 10 mg Torsemide tablet — Single dose 10 mg Torsemide tablet
  Arms: Treatment A; Treatment D
Drug: 25 mg Aldactone (Spironolactone) tablet — Single dose 25 mg Aldactone® (Spironolactone) tablet
  Arms: Treatment B; Treatment D
Drug: FDC (12 mg ER Torsemide + 15mg Spironolactone) tablet — Single dose FDC (12 mg ER Torsemide + 15 mg Spironolactone) tablet
  Arms: Treatment C

SUMMARY:
This study examines the bioavailability and bioequivalence of single dose of a Fixed Dose Combination (FDC) tablet (12 mg Extended-Release Torsemide and 15mg Spironolactone). The goal of this study is to determine PK/PD effects of the FDC, 10 mg Torsemide alone, 25mg Aldactone® (Spironolactone) alone, and 10 mg Torsemide and 25 mg Aldactone® (Spironolactone) taken together in healthy subjects.

DETAILED DESCRIPTION:
Screening and Study Assessments Demographic data, medical, surgical and medication histories, physical examination, height, weight and BMI as well as 12 lead ECG, chest X-ray [PA view], vital signs [blood pressure, pulse rate, respiratory rate and oral temperature], Oxygen Saturation (SpO2 %), hematology, biochemistry, HIV 1 & 2, Hepatitis B and C, RPR test for Syphilis and urinalysis will be done at screening. Females will undergo a serum pregnancy test at the time of screening.

Urine drug screen and breath alcohol test will be done prior to each check-in. Urine pregnancy test will be performed for females prior to each check-in.

Study Duration The total expected study duration is at least 27 days from the day of check-in for Period 1 to the end of Period 4. In case of any post-study laboratory parameter abnormalities, the subject will be followed up at the investigator's discretion.

Washout Period A washout period of at least 07 days will be maintained in between the periods.

Housing Subjects will be housed in the facility from at least 36 hours prior to day of dosing until at least 72 hours post-dose in each period.

Treatments

Treatments Administered:

Treatment (A): 10 mg Torsemide tablet Dose: 1x 10 mg tablet Route of Administration: Oral

Treatment (B): 25 mg Aldactone® (Spironolactone) tablet Dose: 1x 25 mg tablet Route of Administration: Oral

Treatment (C): FDC (12 mg ER Torsemide + 15 mg Spironolactone) tablet. Dose: 1x (12 mg + 15 mg) FDC tablet Route of Administration: Oral

Treatment (D): 10 mg Torsemide tablet and 25 mg Aldactone® (Spironolactone) tablet given together Dose: 1x 10 mg Torsemide tablet + 1x 25 mg Spironolactone tablet Route of Administration: Oral

Blood and Urine Sampling

All subjects will be given a labeled container for urine collection in each period.

Blood samples will be collected in each period.

Adverse and serious adverse events will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

1. Healthy human adult subjects within the age range of 18 to 45 years [both inclusive].
2. Weight not less than 50 kg for male and 45 kg for female and BMI 18.50 to 29.99 kg/m2 [both inclusive].
3. Willingness to provide written informed consent to participate in the study.
4. Subjects should be non-smoker [defined as someone who has stopped smoking for a year before the date of screening] and should not be consuming tobacco containing products.
5. Free of significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
6. Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
7. Subject should be literate.
8. Male subjects must be using two acceptable methods of contraception (e.g., spermicidal gel plus condom) for the entire duration of the study, and upto the study completion visit. Subjects must refrain from fathering a child in the next two weeks following the last study drug administration or have undergone vasectomy (vasectomy must have been done more than 6 months prior to first dosing). Contraceptive usage requirement will be conveyed during the inform consent process. Subjects will be advised to follow effective method of contraception until 2 weeks after the last dose is given.
9. Female subjects of childbearing potential must be using two acceptable methods of contraception, (e.g., intra-uterine device (IUD) plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening and for the duration of the study and for two weeks following the last study drug administration. Contraceptive usage requirement will be conveyed during the inform consent process (or) Postmenopausal women for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy have been performed).

Exclusion Criteria:

Any of the following conditions are cause for exclusion from the study:

1. History or presence of significant: cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, musculoskeletal, psychiatric disease/disorder.
2. History or presence of significance:

   Asthma, urticaria, or other allergic-type reactions after taking Torsemide, Spironolactone or any other drug. Ulceration or history of gastric and/or duodenal ulcer. Stomach or intestinal bleeding. Jaundice in the past 6 months. Internal bleeding.
3. Hypersensitivity or allergy to Torsemide, Spironolactone or any of the excipients.
4. History of alcohol or drug abuse in the past one year.
5. Family history of bleeding disorders.
6. History of difficulty in passing urine or emptying the bladder or of incontinence.
7. Have donated 500 mL or more blood within 90 days before receiving the first dose of the study drug.
8. Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
9. Any difficulty in the accessibility of forearm veins for cannulation or blood sampling and or difficulty with donating blood.
10. Refuse to abstain from food for at least 10 h prior to dosing and for at least 4 h after dosing in each period.
11. Refuse to abstain from fluid for at least 1 h before and 1 h after dosing in each period (except 240 ± 2 mL water given for dosing).
12. Found positive during breath alcohol test done during period one check-in and inability to abstain from alcohol till the end of the study.
13. Found positive during urine drug screening done prior to period one check-in.
14. Found positive screening results for Hepatitis B, Hepatitis C, HIV, or Syphilis.
15. History of difficulty in swallowing tablets.
16. Received any medication [including over-the-counter products], herbal products for 14days preceding the study.
17. Use of enzyme-modifying drugs within 30 days prior to receiving the first dose of study medication.
18. History of dehydration from diarrhea, vomiting, or any other reason within 24 hours prior to check-in of period one.
19. Consumption of xanthine-containing food and beverages (chocolates, tea, coffee, or cola drinks) for at least 48 hours prior to check-in of period one.
20. Consumption of grapefruit or its products within the 48 hours prior to check-in of period one.
21. Female subjects are found to be positive during pregnancy tests done prior to period one check-in.
22. Lactating females.
23. Investigator/Physician feels that it is not in the subject's and/or study's best interest to enroll the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence and bioavailability of the FDC to each of its components | Through study completion: at least 27 days with minimum 7 days washout periods between testing
  Compare bioequivalence and bioavailability (BE and BA) of the FDC to each of the components of the FDC, administered either individually or together: 10 mg Torsemide alone, 25 mg Spironolactone alone and 10 mg Torsemide and 25 mg Spironolactone taken together. Torsemide, Spironolactone, and Canrenone data will be used to estimate the following: Primary pharmacokinetic parameters: Cmax, AUC0-t and AUC0-inf.
Urinary torsemide excretion | Through study completion: at least 27 days with minimum 7 days washout periods between testing
  Urinary torsemide excretion: Rmax, Ae0-24, tmax and percentage drug recovered.

CONTACTS AND LOCATIONS:
Overall Officials: Salim Shah, PhD, JD, Study Chair — Sarfez Pharmaceuticals, Inc.
Locations (1):
- Sarfez Pharmaceuticals, Vienna, Virginia, United States

IPD SHARING:
Plan to Share IPD: No